CLINICAL TRIAL: NCT07363265
Title: A Multicenter, Open-label Phase Ⅱ Study to Evaluate the Efficacy and Safety of LP-005 Injection in Patients With Complement-Mediated Kidney Disease
Brief Title: Efficacy and Safety of LP-005 Injection in Patients With Complement-Mediated Kidney Disease
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Longbio Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P10-LP005-06
Record Dates: First submitted 2026-01-15; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Complement-mediated Renal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LP-005 (Experimental): Patients with complement-mediated renal diseases will be treated with predefined dose of LP-005 (1200 mg or 1500 mg).
  Interventions: Biological: LP-005 Injection

INTERVENTIONS:
Biological: LP-005 Injection — IV, Q4W

SUMMARY:
This is a multicenter, open-label, proof-of-concept, phase Ⅱ adaptive basket clinical trial designed to evaluate the efficacy, safety, and pharmacokinetic profile of LP-005 Injection as add-on therapy to standard treatment in patients with complement-mediated renal diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged 18 to 65 years at screening.
2. Body weight of ≥ 40 kg and a body mass index (BMI) within the range of 15 to 35 kg/m^2 (inclusive).
3. Patients with complement-mediated renal disease.
4. Females and males of childbearing potential (including the participants' partners) must agree to use effective contraceptive measures during the trial and for 3 months after the trial ends.
5. Willing to participate in this clinical trial and voluntarily sign the informed consent form; additionally, be assessed by the investigator as being able to fully understand and comply with all planned study procedures and other requirements.

Exclusion Criteria:

1. Pregnant or lactating female.
2. History of meningococcal infection.
3. Active, uncontrolled acute, chronic, or recurrent infection within 4 weeks prior to screening.
4. Other severe, poorly controlled comorbidities within 3 months prior to screening.
5. Patients with known hypersensitivity to any component of LP-005 or a history of atopic diathesis.
6. History of malignancy within 5 years prior to screening, except for resected cutaneous basal cell carcinoma, resected cutaneous squamous cell carcinoma, and completely resected carcinoma in situ without evidence of local recurrence or metastasis (e.g., cervical carcinoma in situ or breast carcinoma in situ).
7. Prior use of any complement inhibitor within 3 months prior to screening or 5 half-lives of the drug, whichever is longer.
8. Participation in another clinical trial with administration of investigational drug or medical device within 4 weeks prior to screening or 5 half-lives of the administered product, whichever applies.
9. Any condition that, in the investigator's judgment, may impede study participation, pose a safety risk to the participant, or confound the interpretation of study results.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2028-08-02 (Estimated); Study Completion 2029-05-02 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in 24-hour urinary protein-to-creatinine ratio (UPCR) in Basket 1 cohort | Week 24
Proportion of patients with a ≥25% reduction in serum creatinine (SCr) from baseline in Basket 2 cohort | Week 24
Proportion of patients without dialysis requirement in Basket 3 cohort | Week 24

SECONDARY OUTCOMES:
Change from baseline in serum creatinine (SCr) | Up to approximately 64 weeks
Change from baseline in estimated glomerular filtration rate (eGFR) | Up to approximately 64 weeks
Incidence of AEs | Up to approximately 64 weeks
Serum concentrations of LP-005 | Up to approximately 64 weeks
Number of patients with anti-drug antibodies (ADA) | Up to approximately 64 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Minghui Zhao, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, China